CLINICAL TRIAL: NCT02833753
Title: Phase I Trial of Intraperitoneal Oxaliplatin in Combination With Intravenous FOLFIRI (5-fluorouracil, Leucovorin and Irinotecan) for Peritoneal Carcinomatosis From Colorectal and Appendiceal Cancer
Brief Title: Trial of Intraperitoneal (IP) Oxaliplatin in Combination With Intravenous FOLFIRI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Bradley Switzer, Assistant Professor of Medicine, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H00008477
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Cancer; Appendix Cancer; Peritoneal Carcinomatosis
MeSH Terms: conditions — Colorectal Neoplasms; Appendiceal Neoplasms; Peritoneal Neoplasms | interventions — Oxaliplatin

STUDY DESIGN:
Intervention Model Description: There are three cohorts of patients:
  Group #1 is at 25mg/m2 of IP oxaliplatin and has been completed. Group #2 is at 55mg/m2 of IP oxaliplatin is completed. Group #3 is at 85mg/m2 of IP oxaliplatin is currently enrolling. If DLTs found additional 3 subjects will be dosed at the lower dose level cohort.
  2 DLTs were found in the 85 mg/m2 cohort therefore 3 additional subjects (Group # 4) will be enrolled to the 55 mg/m2 cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dose Escalation (Experimental): Single arm dose finding for intraperitoneal Oxaliplatin. All patients will receive experimental treatment.
  The first cohort of 3 patients will receive dose level 1. The second cohort of 3 patients will receive dose level 2. The Third cohort of 3 patients will receive dose level 3. The fourth cohort of 3 patients will receive dose level 2.
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin — Intraperitoneal oxaliplatin will be given along with standard chemotherapy FOLFIRI.
  Level 1: Oxaliplatin 25mg/m2 IP every 2 weeks on day #1 of chemotherapy . Level 2: Oxaliplatin 55mg/m2 IP every 2 weeks on day #1 of chemotherapy Level 3: Oxaliplatin 85mg/m2 IP every 2 weeks on day #1 of chemotherapy Level 4: Oxaliplatin 55 mg/m2 IP every 2 weeks on day #1 of chemotherapy (due to DLTs found)

SUMMARY:
This is a Phase I dose escalation study to determine how much chemotherapy can be safely administered into the abdomen while experiencing the fewest possible side effects.

DETAILED DESCRIPTION:
There are two common combinations of chemotherapy drugs used to treat cancer of the colon, rectum, or appendix that has spread to the abdomen. One uses 5-fluorouracil (also called 5-FU), leucovorin and oxaliplatin, and is called FOLFOX. The other uses 5-FU, leucovorin, and irinotecan, and is called FOLFIRI. The Food and Drug Administration (FDA) has approved each of these combinations as treatment for colon or rectal cancer. Each is given through the veins.

FOLFOX and FOLFIRI do not work well for tumors growing in the abdominal cavity. The investigators are trying to determine if giving chemotherapy called oxaliplatin directly into the abdominal cavity will have a greater effect on the cancer.

The FDA has approved oxaliplatin to be given to people through their veins to treat advanced colorectal cancer. Giving oxaliplatin directly into the abdomen in this study is experimental and is not approved by the FDA. This study will give the standard chemotherapy FOLFIRI through the veins and oxaliplatin directly into the abdomen. This is the first time intraperitoneal oxaliplatin is being given in combination with FOLFIRI.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older and capable of providing informed consent indicating awareness of the investigational nature of this trial, in keeping with institutional policy
* Must consent to participate in the trial and have signed an approved informed consent form conforming to institutional policy
* Must have histopathologically or cytologically confirmed colon, rectal or appendiceal adenocarcinoma with synchronous or metachronous peritoneal dissemination of disease.(Stage IV peritoneal based disease only)
* Must have active measurable disease by either abdominal computerized axial tomography (CT)/ Magnetic resonance imaging (MRI) or laparoscopy.

Adequate laboratory values

* Absolute neutrophil count (ANC) > 1200/10*3/uL
* Platelet count > 140,000/10*3/uL
* Total serum bilirubin ≤ 1.5 mg/dl (patients with total bilirubin >1.5 mg/dL are eligible only with Gilbert's syndrome)
* Alkaline phosphatase < 2.5 times the upper limit of normal (ULN) (alkaline phosphatase and AST cannot both exceed the ULN)
* Aspartate aminotransferase (AST) < 1.5 times the ULN (alkaline phosphatase and AST cannot both exceed the ULN)
* Serum renal function parameters (BUN and creatinine) are within normal limits (eGFR) >50)
* Satisfactory cardiopulmonary function (as determined by Physician)
* Patients can have received prior systemic chemotherapy, radiation or surgery
* Patients must be able to undergo placement of an intraperitoneal (IP) catheter and a Port-A Cath, if not already present
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
* Women of reproductive age and men who are sexually active must be willing to practice effective contraception
* Patients will be allowed to have secondary malignancies as long as they do not require active concomitant treatment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-07; Primary Completion 2022-02 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Define the maximum tolerated dose (MTD) of intraperitoneal (IP) oxaliplatin given with systemic FOLFIRI in patients with peritoneal carcinomatosis (PC) of colorectal or appendiceal origin | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Switzer, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Memorial Medical Center - University Campus, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Falcone A, Ricci S, Brunetti I, Pfanner E, Allegrini G, Barbara C, Crino L, Benedetti G, Evangelista W, Fanchini L, Cortesi E, Picone V, Vitello S, Chiara S, Granetto C, Porcile G, Fioretto L, Orlandini C, Andreuccetti M, Masi G; Gruppo Oncologico Nord Ovest. Phase III trial of infusional fluorouracil, leucovorin, oxaliplatin, and irinotecan (FOLFOXIRI) compared with infusional fluorouracil, leucovorin, and irinotecan (FOLFIRI) as first-line treatment for metastatic colorectal cancer: the Gruppo Oncologico Nord Ovest. J Clin Oncol. 2007 May 1;25(13):1670-6. doi: 10.1200/JCO.2006.09.0928. PMID 17470860
- [Background] Loupakis F, Cremolini C, Masi G, Lonardi S, Zagonel V, Salvatore L, Cortesi E, Tomasello G, Ronzoni M, Spadi R, Zaniboni A, Tonini G, Buonadonna A, Amoroso D, Chiara S, Carlomagno C, Boni C, Allegrini G, Boni L, Falcone A. Initial therapy with FOLFOXIRI and bevacizumab for metastatic colorectal cancer. N Engl J Med. 2014 Oct 23;371(17):1609-18. doi: 10.1056/NEJMoa1403108. PMID 25337750
- [Background] Franko J, Shi Q, Goldman CD, Pockaj BA, Nelson GD, Goldberg RM, Pitot HC, Grothey A, Alberts SR, Sargent DJ. Treatment of colorectal peritoneal carcinomatosis with systemic chemotherapy: a pooled analysis of north central cancer treatment group phase III trials N9741 and N9841. J Clin Oncol. 2012 Jan 20;30(3):263-7. doi: 10.1200/JCO.2011.37.1039. Epub 2011 Dec 12. PMID 22162570
- [Background] Elias D, Lefevre JH, Chevalier J, Brouquet A, Marchal F, Classe JM, Ferron G, Guilloit JM, Meeus P, Goere D, Bonastre J. Complete cytoreductive surgery plus intraperitoneal chemohyperthermia with oxaliplatin for peritoneal carcinomatosis of colorectal origin. J Clin Oncol. 2009 Feb 10;27(5):681-5. doi: 10.1200/JCO.2008.19.7160. Epub 2008 Dec 22. PMID 19103728
- [Background] Sadeghi B, Arvieux C, Glehen O, Beaujard AC, Rivoire M, Baulieux J, Fontaumard E, Brachet A, Caillot JL, Faure JL, Porcheron J, Peix JL, Francois Y, Vignal J, Gilly FN. Peritoneal carcinomatosis from non-gynecologic malignancies: results of the EVOCAPE 1 multicentric prospective study. Cancer. 2000 Jan 15;88(2):358-63. doi: 10.1002/(sici)1097-0142(20000115)88:23.0.co;2-o. PMID 10640968
- [Background] Armstrong DK, Bundy B, Wenzel L, Huang HQ, Baergen R, Lele S, Copeland LJ, Walker JL, Burger RA; Gynecologic Oncology Group. Intraperitoneal cisplatin and paclitaxel in ovarian cancer. N Engl J Med. 2006 Jan 5;354(1):34-43. doi: 10.1056/NEJMoa052985. PMID 16394300
- [Background] Fajardo AD, Tan B, Reddy R, Fleshman J. Delayed repeated intraperitoneal chemotherapy after cytoreductive surgery for colorectal and appendiceal carcinomatosis. Dis Colon Rectum. 2012 Oct;55(10):1044-52. doi: 10.1097/DCR.0b013e318265ad42. PMID 22965403
- [Background] Elias D, Bonnay M, Puizillou JM, Antoun S, Demirdjian S, El OA, Pignon JP, Drouard-Troalen L, Ouellet JF, Ducreux M. Heated intra-operative intraperitoneal oxaliplatin after complete resection of peritoneal carcinomatosis: pharmacokinetics and tissue distribution. Ann Oncol. 2002 Feb;13(2):267-72. doi: 10.1093/annonc/mdf019. PMID 11886004
- [Background] Elias D, Matsuhisa T, Sideris L, Liberale G, Drouard-Troalen L, Raynard B, Pocard M, Puizillou JM, Billard V, Bourget P, Ducreux M. Heated intra-operative intraperitoneal oxaliplatin plus irinotecan after complete resection of peritoneal carcinomatosis: pharmacokinetics, tissue distribution and tolerance. Ann Oncol. 2004 Oct;15(10):1558-65. doi: 10.1093/annonc/mdh398. PMID 15367418
- [Background] Gervais MK, Dube P, McConnell Y, Drolet P, Mitchell A, Sideris L. Cytoreductive surgery plus hyperthermic intraperitoneal chemotherapy with oxaliplatin for peritoneal carcinomatosis arising from colorectal cancer. J Surg Oncol. 2013 Dec;108(7):438-43. doi: 10.1002/jso.23431. Epub 2013 Sep 9. PMID 24018983
- [Background] Ceelen W, De Somer F, Van Nieuwenhove Y, Vande Putte D, Pattyn P. Effect of perfusion temperature on glucose and electrolyte transport during hyperthermic intraperitoneal chemoperfusion (HIPEC) with oxaliplatin. Eur J Surg Oncol. 2013 Jul;39(7):754-9. doi: 10.1016/j.ejso.2012.07.120. Epub 2012 Aug 9. PMID 22878060
- [Background] Mehta AM, Van den Hoven JM, Rosing H, Hillebrand MJ, Nuijen B, Huitema AD, Beijnen JH, Verwaal VJ. Stability of oxaliplatin in chloride-containing carrier solutions used in hyperthermic intraperitoneal chemotherapy. Int J Pharm. 2015 Feb 1;479(1):23-7. doi: 10.1016/j.ijpharm.2014.12.025. Epub 2014 Dec 20. PMID 25535649
- [Background] Fuchs CS, Marshall J, Mitchell E, Wierzbicki R, Ganju V, Jeffery M, Schulz J, Richards D, Soufi-Mahjoubi R, Wang B, Barrueco J. Randomized, controlled trial of irinotecan plus infusional, bolus, or oral fluoropyrimidines in first-line treatment of metastatic colorectal cancer: results from the BICC-C Study. J Clin Oncol. 2007 Oct 20;25(30):4779-86. doi: 10.1200/JCO.2007.11.3357. PMID 17947725
- [Background] Teefey P, Bou Zgheib N, Apte SM, Gonzalez-Bosquet J, Judson PL, Roberts WS, Lancaster JM, Wenham RM. Factors associated with improved toxicity and tolerability of intraperitoneal chemotherapy in advanced-stage epithelial ovarian cancers. Am J Obstet Gynecol. 2013 Jun;208(6):501.e1-7. doi: 10.1016/j.ajog.2013.03.012. Epub 2013 Mar 15. PMID 23507546
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774